CLINICAL TRIAL: NCT05754931
Title: Effects of Deep Neck Flexors Training Versus Muscle Energy Technique on Cervicogenic Headache
Brief Title: Deep Neck Flexors Training Versus Muscle Energy Technique on Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hirah Naseem
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Cervicogenic Headache
Keywords: Cervicogenic Headache; Neck Muscles; exercise muscle stretch; postures
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deep neck flexor group (Experimental): Deep neck flexors stretch
  Conventional Therapy:
  Moist heat therapy for 10 minutes, TENS 10 min, cervical active ROMS, Non-thrust mobilizations
  Interventions: Other: Deep neck flexors training + Conventional therapy
- muscle energy technique (Active Comparator): Post isometric stretch on trapezious and suboccipital muscles
  Conventional Therapy:
  Moist heat therapy for 10 minutes, TENS 10 min, cervical active ROMS, Non-thrust mobilizations
  Interventions: Other: Muscles energy techniques + conventional therapy

INTERVENTIONS:
Other: Deep neck flexors training + Conventional therapy — Hold for 10 sec and repeated 10 times.Patients will be treated 3 times a week for 4 consecutive weeks
  Arms: deep neck flexor group
Other: Muscles energy techniques + conventional therapy — position of patient is in maximal comfort and lengthening After engaging the barrier use of an isometric contraction Feel the release and lengthen the muscle repeated for 4 time per session Patients will be treated 3 times a week for 4 consecutive weeks
  Arms: muscle energy technique

SUMMARY:
Aim of this study is to compare the effects of deep neck flexors stretching versus muscles energy technique on pain, cervical range of motion, sleep disturbance and cervical spine posture in patients with Cervicogenic headache and interpret which technique is better among both.A randomized control trial that will include total 28 participants.The first group will receive deep neck flexors stretching along with conventional therapy and 2nd group will receive muscles energy technique along with conventional therapy.Data collected will be analyzed through SPSS 25.

DETAILED DESCRIPTION:
Cervicogenic headache is a disabling condition associated with musculoskeletal impairment of the cervical region.Cervicogenic headache is a clinical syndrome characterized by primarily unilateral pain that originates in the neck, typically provoked by neck movement or pressure over tender points in the neck, with reduced range of movement of the cervical spine.Cervicogenic Headache is pain referred to the head from a source in the cervical spine. It can influence the patient's quality of life in addition to a loss of functions when compared with the groups with other headache disorders.

A variety of invasive and noninvasive therapeutic modalities are used in the treatment of cervicogenic headache.Physical therapy is considered as most effective treatment of cervicogenic headache including modalities, manual therapy, muscle stretching, Muscle Energy Techniques, deep neck flexors training, Instrument-Assisted Soft Tissue Mobilization , therapeutic exercises and kinesiology tapping.Deep cervical flexor exercise is a low-load exercise focused on deep cervical flexor muscles, as described by Jull et al. This exercise targets the deep flexor muscles of the cervical region, rather than the superficial flexor muscles. Deep neck flexor training is said to improve the Cervicogenic headache according to the literature review.

According to the Literature review, in cervicogenic headache 2 group of muscles are involved i.e. deep cervical flexors (longus colli, longus capitis, Rectus capitis and Longus capitus) gets weakened and cervical extensors (suboccipital and upper trapezius) gets tightened. It is evident that deep neck flexor training is effective in improving pain, cervical range of motion and posture in Cervicogenic headache. Muscle Energy techniques are also proven to reduce pain and improve range of motion so post isometric relaxation will use in this study. Limited literature is available which compares the effects of post isometric relaxation deep neck flexors and specifically on Cervicogenic headaches. Aim of this study is to compare the effects of these techniques on pain, cervical range of motion, sleep disturbance and cervical spine posture in patients with Cervicogenic headache and interpret which technique is better among both. I hope that this study will add valuable literature and scope for future researchers to work on this topic.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 - 55 years.
* Both male and female subjects will be recruited in the study.
* Unilateral headache (without side shift) related by pain, movement and sustaining
* position of neck started from the occiput spread to the tempro-frontal region for more than 3 months
* >20 degree movement restriction in cervical ROM, especially in the upper cervical rotation.
* Positive flexion rotation test to confirm Cervicogenic headache.
* Subjects with rounded shoulders having distance between on the table and the acromion>2.5 cm

Exclusion Criteria:

* Fracture or previous surgery on vertebral column
* History of spinal stenosis or disc prolapse
* dysfunction or headache with autonomic involvement
* Other types of headache including migraine, tension type etc.
* laxity of alar ligaments
* vertebra basilar artery insufficiency
* Patients with a history of physiotherapy at least 3 months prior to the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain rating scale | 4 weeks
  The Numeric Pain Rating Scale (NPRS) measures the subjective intensity of pain.

SECONDARY OUTCOMES:
Inclinometer | 4 weeks
  Measurements of cervical flexion, extension, lateral flexion, and rotation will be measured using inclinometer
Cervical posture | 4 weeks
  For measurement of cervical posture, photographs taken from the side were used for objective measurement of forward head posture
Insomnia Severity Index (ISI) | 4 weeks
  It is a brief self-report questionnaire that measures the patient's perception of insomnia severity

CONTACTS AND LOCATIONS:
Overall Officials: Madiha Ali, MSOPMT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No